CLINICAL TRIAL: NCT05402215
Title: The Effect of the Flipped Classroom Model on Teaching Clinical Practice Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali Kaplan, Lecturer Dr., TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: TC Kayseri University
Record Dates: First submitted 2022-05-30; First posted 2022-06-02 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Flipped Classroom Model in Teaching
Keywords: Flipped classroom model; Clinical Practice Skills; Nursing
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: stratified randomization method
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The flipped classroom model was used in teaching the clinical practice skills of the students in the experimental group. First of all, videos for clinical applications were prepared by the researchers. These prepared videos were shared with the students in the experimental group one week before the lesson day of each application for preliminary study and the students were asked to work on these videos. On the day of the lesson, group work, question-answer and discussion activities were held with the students in the classroom environment. At the end of the lesson, the students were asked to do the applications on the simulation models of the application and the checklists were filled.
  Interventions: Behavioral: The flipped classroom model was used to teach students' clinical practice skills.
- control group (Active Comparator): To the students in the control group, the application was explained by the researcher (instructor conducting the course) using presentation and demonstration methods. Each application was made on different days. The prepared checklists were filled by the other researcher. While the students were doing the applications, one of the researchers observed the application and marked only the skill level in the checklists ("applied", "incompletely applied" and "did not apply") without making any comments or directions.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: The flipped classroom model was used to teach students' clinical practice skills. — Videos for clinical applications have been prepared by researchers. These prepared videos were shared with the students in the experimental group one week before the lesson day of each application for preliminary study and the students were asked to work on these videos. On the day of the lesson, group work, question-answer and discussion activities were held with the students in the classroom environment. At the end of the lesson, the students were asked to do the applications on the simulation models of the application and the checklists were filled.
  Arms: experimental group
Behavioral: control group — To the students in the control group, the application was explained by the researcher (instructor conducting the course) using presentation and demonstration methods. Each application was made on different days. The prepared checklists were filled by the other researcher.
  Arms: control group

SUMMARY:
This research is a randomized controlled experimental study planned to examine the effect of the flipped classroom model in teaching clinical practice skills. The research was carried out on first year students of the First and Emergency Aid Program at a state university in Turkey. The data were collected for one year, in the fall and spring terms. The universe of the research consisted of 46 students enrolled in the 2021-2022 Academic Year First and Emergency Aid Program and studying in the first year. In the study, stratified randomization method was used since it was thought that random selection could affect the study statistically in assigning students to groups. The data of the study were collected using the "Descriptive Characteristics Information Form", which includes the introductory information of the students, and the "Check List", which includes the clinical practice skill steps. While the flipped classroom model was used in teaching clinical practice skills of students in the experimental group, standard lectures were used in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old

Exclusion Criteria:

* who refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

PRIMARY OUTCOMES:
Control List | immediately after application
  The checklists were created by the researchers using the clinical practice guidelines on nursing principles (Dikmen & Akın Korhan, 2016; Taşçı, et al., 2018) and the opinions of three experts in the field of nursing principles were obtained. In the study, intravenous catheterization (28 application steps), intravenous blood collection (24 application steps), blood pressure measurement from the brachial artery (24 application steps), intramuscular injection into the ventrogluteal region (34 application steps) and female urinary catheterization (39 application steps) applications were examined. 5 checklists containing skill steps were used. In the checklists, each application step was arranged as a three-point Likert scale as "applied" (2 points), "applied incompletely" (1 point), and "did not apply" (0 points). The lowest score in the checklists is 0, and the highest score differs according to the number of skill steps in clinical applications.

CONTACTS AND LOCATIONS:
Overall Officials: Ali KAPLAN, Dr., Principal Investigator — Kayseri University
Locations (1):
- Kayseri Üniversitesi, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No